CLINICAL TRIAL: NCT04485325
Title: Capability of Tofacitinib or Etanercept to Accelerate Clinical Relevant Tapering of Non-steroidal Anti-inflammatory Drugs (NSAID) and Treat-to-target Guided De-escalation of Corticosteroids in Patients With Active Rheumatoid Arthritis (RA) and an Inadequate Response to Previous csDMARD Therapy (AcceleRAte)
Brief Title: Capability of Tofacitinib or Etanercept to Accelerate Tapering of NSAID and Treat-to-target Guided De-escalation of Corticosteroids in RA Patients
Acronym: AcceleRAte
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Frank Behrens (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Dr. Frank Behrens, Representative of the Sponsor, Fraunhofer Institute for Translational Medicine and Pharmacology ITMP
Organization: Fraunhofer Institute for Translational Medicine and Pharmacology ITMP (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMP-0731-2018
Record Dates: First submitted 2020-04-30; First posted 2020-07-24 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Rheumatic Arthritis
Keywords: treat-to-target; pain
MeSH Terms: conditions — Rheumatic Fever; Pain | interventions — tofacitinib; 5-(tetradecyloxy)-2-furancarboxylic acid; Etanercept; Receptor, Endothelin A

STUDY DESIGN:
Intervention Model Description: two arm, randomized, open-label, parallel group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tofacitinib (Active Comparator): Tofacitinib (Xeljanz®; 5 mg twice daily, p.o.)
  Interventions: Drug: Tofacitinib
- Etanercept (Active Comparator): Etanercept (Enbrel®; 50 mg once per week, s.c.)
  Interventions: Biological: Etanercept

INTERVENTIONS:
Drug: Tofacitinib — 5 mg twice daily, p.o.
  Other Names: TOFA, Xeljanz
  Arms: Tofacitinib
Biological: Etanercept — 50 mg once per week, s.c.
  Other Names: Enbrel, ETA
  Arms: Etanercept

SUMMARY:
Patients with active rheumatic arthritis (RA) and lack of efficacy of at least one csDMARD (Disease-modifying anti-rheumatic drug) treatment will be randomized to receive either Tofacitinib (TOFA) or etanercept (ETA). The study will be separated into two parts: The capability to decrease and discontinue pain-reducing treatment with a NSAID (non-steroidal anti-inflammatory drug) over the first 12 weeks of treatment will be measured for primary outcome measured using a visual analogue scale (VAS) at week 12 compared to baseline between the two treatment groups.

Starting at week 12, the capability to taper corticosteroid (CS) treatment using a treat-to-target strategy, i.e. when at least low disease activity (LDA-DAS28) is achieved, will be measured in both groups.

DETAILED DESCRIPTION:
In this clinical study, a design was chosen to reflect European standards recommended by EULAR for treatment of active RA by comparison of a Treat-to- target (T2T) approach in two treatment groups: Patients with active RA and lack of efficacy of at least one csDMARD treatment will be randomized to receive either TOFA or ETA. The study will be separated into two parts: The capability to decrease and discontinue pain-reducing treatment with a NSAID (Celecoxib, two times 200 mg as maximum standard dosage for RA) over the first 12 weeks of treatment will be measured for primary outcome. The proportion of patients with successful discontinuation of Celecoxib and significant and clinical relevant decrease of pain-levels measured using a visual analogue scale (VAS) with a reduction of at least 30% at week 12 compared to baseline will be compared between the two treatment groups.

Starting at week 12, the capability to taper CS treatment using a treat-to-target strategy, i.e. when at least low disease activity (LDA-DAS28) is achieved, will be measured in both groups. In addition to efficacy assessments (DAS28, ACR-response, SJC, TJC), patient reported outcomes, Quality of Life (QoL) measurements and patient satisfaction will be evaluated. Safety (severity and frequency of adverse events) will be evaluated over the 24-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active RA and an inadequate response to up to two previous conventional synthetic Disease modifying anti-rheumatic drug (csDMARD) treatments (methotrexate (MTX), leflunomide (LEF),sulfasalazine (SSZ)) with or without ongoing csDMARD therapy
* RA according to ACR classification criteria
* Age 18 - 65 years
* Active RA is defined as

  * DAS28 > 3.2 and
  * TJC ≥ 3 and SJC ≥ 3
* VAS-pain ≥ 60 mm (0-100 mm)
* Accompanying CS treatment for RA with a stable dosage of ≥ 2mg/d and ≤ 10 mg/d 2 weeks prior to BL (not more than 30% of patients without CS)
* Accompanying need of NSAID or analgesic treatment due to arthritis and in dosages not exceeding the maximum dose according to Summary of Product characteristics (SmPC)
* If ongoing csDMARD treatment, stable treatment will be defined as either

  * MTX treatment with a dosage of ≥ 10 mg/week and ≤ 25 mg/week, continuously for at least 12 weeks prior to Screening (SCR) with a stable dose of MTX for at least 2 weeks prior to BL or
  * LEF treatment with a dosage between 10 to 20 mg/day, continuously for at least 12 weeks prior to SCR with a stable dose of LEF for at least 2 weeks prior to BL or
  * SSZ treatment with dosage between 1 to 3 g/day, continuously for at least 12 weeks prior to SCR with a stable dose of SSZ for at least 2 weeks prior to BL
* Presence of documented negative results for testing of Hepatitis B and C
* Completed SARS-CoV-2-immunisation as currently recommended by the Standing Committee of Vaccination
* Written informed consent obtained prior to the initiation of any protocol-required procedures
* Willingness to comply to study procedures and study protocol

Exclusion Criteria:

* Previous use of Tofacitinib or other Janus-Kinase (JAK)-inhibitors
* Previous use of Etanercept
* Previous use of any biological agent for RA

  * which was stopped due to lack of efficacy
  * one previous use of biological stopped due to intolerance will be allowed
* CS treatment with dosages >10 mg at BL
* Known hypersensitivity to any component of the study medication (TOFA, ETA, Celecoxib)
* Previous use of Celecoxib as analgesic therapy which was stopped due to lack of efficacy or intolerance
* Concomitant diseases with chronic pain syndrome or need of extended dosages or long-term treatment with the maximum dosages of NSAID/analgesics (according to SmPC) due to other concomitant diseases/pain symptoms in discretion of the treating physician Exclusion criteria related to general health
* Patients with other chronic inflammatory articular disease or systemic autoimmune disease
* Patients with active Tuberculosis (Tb) (evaluation of Tb according to local standards in clinical care)
* Patients with latent Tb, that are not pre-treated for at least 1 month and planned to be treated 9 months in total with Isozid once a day
* Any active infection, a history of recurrent clinically significant infections (e.g. human immune deficiency virus (HIV)), or a history of recurrent bacterial infections with encapsulated organisms
* Primary or secondary immunodeficiency
* Current malignancy or history of malignancies except adequately treated or excised basal cell or squamous cell carcinoma or cervical carcinoma in situ.
* Patients of 50 years and older, if they have one or more cardiovascular risk factors (CVRF) defined as:

  * Current cigarette smoking,
  * Known diagnosis of hypertension,
  * HDL <40 mg/dl,
  * Diabetes mellitus,
  * History of coronary artery disease: history of revascularization procedure, coronary artery bypass grafting, myocardial infarction, cardiac arrest, unstable angina, acute coronary syndrome or
  * History of premature coronary heart disease or sudden death documented in first degree relatives (male relative before 55 years, female relative before 65 years)
* Evidence of significant uncontrolled concomitant diseases or serious and/or uncontrolled diseases that are likely to interfere with the evaluation of the patient's safety and with the study outcome
* History of a severe psychological illness or condition
* Known hypersensitivity to sulfonamides
* Active peptic ulceration or gastrointestinal (GI) bleeding
* Patients who have experienced asthma, acute rhinitis, nasal polyps, angioneurotic oedema, urticaria or other allergic-type reactions after taking acetylsalicylic acid (aspirin) or other NSAIDs including Cyclooxigenase (COX)-2 inhibitors
* Risk for or history of thrombotic events (e.g. pulmonary embolism or thrombosis) Severe hepatic dysfunction (serum albumin < 25 g/L or Child-Pugh score ≥ 10)
* Patients with estimated creatinine clearance < 30 mL/min
* Inflammatory bowel disease
* Congestive heart failure (New York Heart Association (NYHA) II-IV)
* Established ischaemic heart disease, peripheral arterial disease and/or cerebrovascular disease
* Women lactating, pregnant, nursing or of childbearing potential with a positive pregnancy test
* Males or females of reproductive potential not willing to use effective contraception (e.g. contraceptive pill, intrauterine device (IUD), physical barrier)
* Alcohol, drug or chemical abuse Exclusion criteria related to prior treatments
* Current participation in another interventional clinical trial or participation within the last 90 days Exclusion criteria related to formal aspects
* Underage or incapable patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Discontinuation of Celecoxib treatment and clinically relevant improvement in pain | Baseline to week 12
  Proportion of patients who can discontinue Celecoxib treatment and in whom clinically relevant improvement in pain levels are measured, defined as reduction in VAS pain of ≥ 30%

SECONDARY OUTCOMES:
Mean dosage of Celecoxib in patients | at 12 weeks
  Mean dosage of Celecoxib in patients
discontinuation of CS-treatment | at week 24
  Proportion of patients with discontinuation of CS-treatment at week 24
rescue treatment | at week 12
  Proportion of patients who require rescue treatment at week 12
Mean dosage of Corticosteroids (CS) in the patients who achieve Low Disease activity (LDA) in the two treatment groups | at week 24
  Mean dosage of CS in the patients who achieve LDA at week 24 in the two treatment groups
Mean dosage of Corticosteroids (CS) | at week 24
  Mean dosage of CS at week 24 (W24)
NSAID treatment | at week 24
  Number of patients with NSAID treatment at W24
re-started NSAID treatment | week 12 to week 24
  Proportion of patients who re-started NSAID treatment after week 12 (W12) until W24
Absolute pain levels | at week 2
  Absolute pain levels measured by visual analogue scale (VAS). minimum is 0 mm, maximum is 100 mm whereas 0 is no pain and 100 is worst
Absolute pain levels | at week 4
  Absolute pain levels measured by visual analogue scale (VAS). minimum is 0 mm, maximum is 100 mm whereas 0 is no pain and 100 is worst
Absolute pain levels | at week 8
  Absolute pain levels measured by visual analogue scale (VAS). minimum is 0 mm, maximum is 100 mm whereas 0 is no pain and 100 is worst
Absolute pain levels | at week 12
  Absolute pain levels measured by visual analogue scale (VAS). minimum is 0 mm, maximum is 100 mm whereas 0 is no pain and 100 is worst
Absolute pain levels | at week 16
  Absolute pain levels measured by visual analogue scale (VAS). minimum is 0 mm, maximum is 100 mm whereas 0 is no pain and 100 is worst
Absolute pain levels | at week 20
  Absolute pain levels measured by visual analogue scale (VAS). minimum is 0 mm, maximum is 100 mm whereas 0 is no pain and 100 is worst
Absolute pain levels | at week 24
  Absolute pain levels measured by visual analogue scale (VAS). minimum is 0 mm, maximum is 100 mm whereas 0 is no pain and 100 is worst
relative (percent) pain levels | at week 2
  relative (percent) pain levels measured by visual analogue scale (VAS). minimum is 0 mm, maximum is 100 mm whereas 0 is no pain and 100 is worst
relative (percent) pain levels | at week 4
  relative (percent) pain levels measured by visual analogue scale (VAS). minimum is 0 mm, maximum is 100 mm whereas 0 is no pain and 100 is worst
relative (percent) pain levels | at week 8
  relative (percent) pain levels measured by visual analogue scale (VAS). minimum is 0 mm, maximum is 100 mm whereas 0 is no pain and 100 is worst
relative (percent) pain levels | at week 12
  relative (percent) pain levels measured by visual analogue scale (VAS). minimum is 0 mm, maximum is 100 mm whereas 0 is no pain and 100 is worst
relative (percent) pain levels | at week 16
  relative (percent) pain levels measured by visual analogue scale (VAS). minimum is 0 mm, maximum is 100 mm whereas 0 is no pain and 100 is worst
relative (percent) pain levels | at week 20
  relative (percent) pain levels measured by visual analogue scale (VAS). minimum is 0 mm, maximum is 100 mm whereas 0 is no pain and 100 is worst
relative (percent) pain levels | at week 24
  relative (percent) pain levels measured by visual analogue scale (VAS). minimum is 0 mm, maximum is 100 mm whereas 0 is no pain and 100 is worst
Change in pain levels | at week 2
  Change in pain levels measured by visual analogue scale (VAS) compared to BL. minimum is 0 mm, maximum is 100 mm whereas 0 is no pain and 100 is worst
Change in pain levels | at week 4
  Change in pain levels visual analogue scale (VAS) compared to BL. minimum is 0 mm, maximum is 100 mm whereas 0 is no pain and 100 is worst
Change in pain levels | at week 8
  Change in pain levels visual analogue scale (VAS) compared to BL. minimum is 0 mm, maximum is 100 mm whereas 0 is no pain and 100 is worst
Change in pain levels | at week 12
  Change in pain levels visual analogue scale (VAS) compared to BL. minimum is 0 mm, maximum is 100 mm whereas 0 is no pain and 100 is worst
Change in pain levels | at week 16
  Change in pain levels visual analogue scale (VAS) compared to BL. minimum is 0 mm, maximum is 100 mm whereas 0 is no pain and 100 is worst
Change in pain levels | at week 20
  Change in pain levels visual analogue scale (VAS) compared to BL. minimum is 0 mm, maximum is 100 mm whereas 0 is no pain and 100 is worst
Change in pain levels | at week 24
  Change in pain levels visual analogue scale (VAS) compared to BL. minimum is 0 mm, maximum is 100 mm whereas 0 is no pain and 100 is worst
Determination of flares | between week 12 and week 24
  Determination of flares (measured by FLARE questionnaire) between week 12 and week 24
Proportion of LDA | at week 4
  Proportion of patients who achieve LDA (Disease Activity Score 28 (DAS28) calculated by Erythrocyte sediment rate (ESR) (DAS28 (ESR) ≤ 3.2)
Proportion of LDA | at week 12
  Proportion of patients who achieve LDA (Disease Activity Score 28 (DAS28) calculated by Erythrocyte sediment rate (ESR) (DAS28 (ESR) ≤ 3.2)
Proportion of LDA | at week 16
  Proportion of patients who achieve LDA (Disease Activity Score 28 (DAS28) calculated by Erythrocyte sediment rate (ESR) (DAS28 (ESR) ≤ 3.2)
Proportion of LDA | at week 20
  Proportion of patients who achieve LDA (Disease Activity Score 28 (DAS28) calculated by Erythrocyte sediment rate (ESR) (DAS28 (ESR) ≤ 3.2)
Proportion of LDA | at week 24
  Proportion of patients who achieve LDA (Disease Activity Score 28 (DAS28) calculated by Erythrocyte sediment rate (ESR) (DAS28 (ESR) ≤ 3.2)
Proportion of DAS remission | at week 4
  Proportion of patients who achieve DASremission (Disease Activity Score 28 (DAS28) calculated by Erythrocyte sediment rate (ESR) DAS28 (ESR) ≤ 2.6)
Proportion of DAS remission | at week 12
  Proportion of patients who achieve DASremission (Disease Activity Score 28 (DAS28) calculated by Erythrocyte sediment rate (ESR) DAS28 (ESR) ≤ 2.6)
Proportion of DAS remission | at week 16
  Proportion of patients who achieve DASremission (Disease Activity Score 28 (DAS28) calculated by Erythrocyte sediment rate (ESR) DAS28 (ESR) ≤ 2.6)
Proportion of DAS remission | at week 20
  Proportion of patients who achieve DASremission (Disease Activity Score 28 (DAS28) calculated by Erythrocyte sediment rate (ESR) DAS28 (ESR) ≤ 2.6)
Proportion of DAS remission | at week 24
  Proportion of patients who achieve DASremission (Disease Activity Score 28 (DAS28) calculated by Erythrocyte sediment rate (ESR) DAS28 (ESR) ≤ 2.6)
Proportion of ACR20 response | at week 4
  Proportion of patients who achieve ACR20 response - measure based on American College of Rheumatology (ACR) criteria improvement of at least 20%
Proportion of ACR20 response | at week 12
  Proportion of patients who achieve ACR20 response - measure based on American College of Rheumatology (ACR) criteria improvement of at least 20%
Proportion of ACR20 response | at week 16
  Proportion of patients who achieve ACR20 response - measure based on American College of Rheumatology (ACR) criteria improvement of at least 20%
Proportion of ACR20 response | at week 20
  Proportion of patients who achieve ACR20 response - measure based on American College of Rheumatology (ACR) criteria improvement of at least 20%
Proportion of ACR20 response | at week 24
  Proportion of patients who achieve ACR20 response - measure based on American College of Rheumatology (ACR) criteria improvement of at least 20%
Proportion of ACR 50 response | at week 4
  Proportion of patients who achieve ACR50 response - measure based on American College of Rheumatology (ACR) criteria improvement of at least 50%
Proportion of ACR 50 response | at week 12
  Proportion of patients who achieve ACR50 response - measure based on American College of Rheumatology (ACR) criteria improvement of at least 50%
Proportion of ACR 50 response | at week 16
  Proportion of patients who achieve ACR50 response - measure based on American College of Rheumatology (ACR) criteria improvement of at least 50%
Proportion of ACR 50 response | at week 20
  Proportion of patients who achieve ACR50 response - measure based on American College of Rheumatology (ACR) criteria improvement of at least 50%
Proportion of ACR 50 response | at week 24
  Proportion of patients who achieve ACR50 response - measure based on American College of Rheumatology (ACR) criteria improvement of at least 50%
Proportion of ACR 70 response | at week 4
  Proportion of patients who achieve ACR70 response - measure based on American College of Rheumatology (ACR) criteria improvement of at least 70%
Proportion of ACR 70 response | at week 12
  Proportion of patients who achieve ACR70 response - measure based on American College of Rheumatology (ACR) criteria improvement of at least 70%
Proportion of ACR 70 response | at week 16
  Proportion of patients who achieve ACR70 response - measure based on American College of Rheumatology (ACR) criteria improvement of at least 70%
Proportion of ACR 70 response | at week 20
  Proportion of patients who achieve ACR70 response - measure based on American College of Rheumatology (ACR) criteria improvement of at least 70%
Proportion of ACR 70 response | at week 24
  Proportion of patients who achieve ACR70 response - measure based on American College of Rheumatology (ACR) criteria improvement of at least 70%
Changes in ACR core set | at baseline
  Changes in ACR core set
Changes in ACR core set | at week 4
  Changes in ACR core set
Changes in ACR core set | at week 12
  Changes in ACR core set
Changes in ACR core set | at week 16
  Changes in ACR core set
Changes in ACR core set | at week 20
  Changes in ACR core set
Changes in ACR core set | at week 24
  Changes in ACR core set change
DAS28 (ESR) | at baseline
  DAS28 (ESR) change compared to BL
DAS28 (ESR) | at week 4
  DAS28 (ESR) change compared to BL
DAS28 (ESR) | at week 12
  DAS28 (ESR) change compared to BL
DAS28 (ESR) | at week 16
  DAS28 (ESR) change compared to BL
DAS28 (ESR) | at week 20
  DAS28 (ESR) change compared to BL
DAS28 (ESR) | at week 24
  DAS28 (ESR) change compared to BL
SJC (66), | at baseline
  Swollen joint count (66 joints) change compared to BL
SJC (66), | at week 4
  Swollen joint count (66 joints) change compared to BL
SJC (66), | at week 12
  Swollen joint count (66 joints) change compared to BL
SJC (66), | at week 16
  Swollen joint count (66 joints) change compared to BL
SJC (66), | at week 20
  Swollen joint count (66 joints) change compared to BL
SJC (66), | at week 24
  Swollen joint count (SJC) (66 joints) change compared to BL
TJC (68) | at baseline
  tender joint count (TJC) - 68 joints change compared to BL
TJC (68) | at week 4
  tender joint count (TJC) - 68 joints change compared to BL
TJC (68) | at week 12
  tender joint count (TJC) - 68 joints change compared to BL
TJC (68) | at week 16
  tender joint count (TJC) - 68 joints change compared to BL
TJC (68) | at week 20
  tender joint count (TJC) - 68 joints change compared to BL
TJC (68) | at week 24
  tender joint count (TJC) - 68 joints change compared to BL
Quality of Life: SF36 (36 items short form health survey) | at baseline
  Quality of Life: SF36 scores
Quality of Life: SF36 (36 items short form health survey) | at week 4
  Quality of Life: SF36 scores.SF36 is a 36 items short form health survey and consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Change in Quality of Life: SF36 (36 items short form health survey) | at week 4
  Quality of Life: SF36 change to BL. SF36 is a 36 items short form health survey and consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Quality of Life: SF36 (36 items short form health survey) | at week 12
  Quality of Life: SF36 scores. SF36 is a 36 items short form health survey and consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Change in Quality of Life: SF36 (36 items short form health survey) | at week 12
  Quality of Life: SF36 change to BL. SF36 is a 36 items short form health survey and consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Quality of Life: SF36 (36 items short form health survey) | at week 16
  Quality of Life: SF36 scores. SF36 is a 36 items short form health survey and consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Change in Quality of Life: SF36 (36 items short form health survey) | at week 16
  Quality of Life: SF36 change to BL. SF36 is a 36 items short form health survey and consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Quality of Life: SF36 (36 items short form health survey) | at week 20
  Quality of Life: SF36 scores. SF36 is a 36 items short form health survey and consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Change in Quality of Life: SF36 (36 items short form health survey) | at week 20
  Quality of Life: SF36 change to BL. SF36 is a 36 items short form health survey and consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Quality of Life: SF36 (36 items short form health survey) | at week 24
  Quality of Life: SF36 scores. SF36 is a 36 items short form health survey and consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Change in Quality of Life: SF36 (36 items short form health survey) | at week 24
  Quality of Life: SF36 change to BL. SF36 is a 36 items short form health survey and consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Quality of Life HAQ-DI (health assessment questionnaire - disability index) | at baseline
  Quality of Life HAQ-DI scores The HAQ-DI is a health assessment questionnaire - disability index that consists of 8 subcategories. For each the single scales range from 0 (no difficulty) to 3 (unable to do).
Quality of Life HAQ-DI (health assessment questionnaire - disability index) | at week 4
  Quality of Life HAQ-DI scores. The HAQ-DI is a health assessment questionnaire - disability index that consists of 8 subcategories. For each the single scales range from 0 (no difficulty) to 3 (unable to do).
Change in Quality of Life HAQ-DI (health assessment questionnaire - disability index) | at week 4
  Quality of Life HAQ-DI change to BL. The HAQ-DI is a health assessment questionnaire - disability index that consists of 8 subcategories. For each the single scales range from 0 (no difficulty) to 3 (unable to do).
Quality of Life HAQ-DI (health assessment questionnaire - disability index) | at week 12
  Quality of Life HAQ-DI scores. The HAQ-DI is a health assessment questionnaire - disability index that consists of 8 subcategories. For each the single scales range from 0 (no difficulty) to 3 (unable to do).
Change of Quality of Life HAQ-DI (health assessment questionnaire - disability index) | at week 12
  Quality of Life HAQ-DI change to BL. The HAQ-DI is a health assessment questionnaire - disability index that consists of 8 subcategories. For each the single scales range from 0 (no difficulty) to 3 (unable to do).
Quality of Life HAQ-DI (health assessment questionnaire - disability index) | at week 16
  Quality of Life HAQ-DI scores. The HAQ-DI is a health assessment questionnaire - disability index that consists of 8 subcategories. For each the single scales range from 0 (no difficulty) to 3 (unable to do).
Change of Quality of Life HAQ-DI (health assessment questionnaire - disability index) | at week 16
  Quality of Life HAQ-DI change to BL. The HAQ-DI is a health assessment questionnaire - disability index that consists of 8 subcategories. For each the single scales range from 0 (no difficulty) to 3 (unable to do).
Quality of Life HAQ-DI (health assessment questionnaire - disability index) | at week 20
  Quality of Life HAQ-DI scores.The HAQ-DI is a health assessment questionnaire - disability index that consists of 8 subcategories. For each the single scales range from 0 (no difficulty) to 3 (unable to do).
Change of Quality of Life HAQ-DI (health assessment questionnaire - disability index) | at week 20
  Quality of Life HAQ-DI change to BL. The HAQ-DI is a health assessment questionnaire - disability index that consists of 8 subcategories. For each the single scales range from 0 (no difficulty) to 3 (unable to do).
Quality of Life HAQ-DI (health assessment questionnaire - disability index) | at week 24
  Quality of Life HAQ-DI scores. The HAQ-DI is a health assessment questionnaire - disability index that consists of 8 subcategories. For each the single scales range from 0 (no difficulty) to 3 (unable to do).
Change of Quality of Life HAQ-DI (health assessment questionnaire - disability index) | at week 24
  Quality of Life HAQ-DI change to BL. The HAQ-DI is a health assessment questionnaire - disability index that consists of 8 subcategories. For each the single scales range from 0 (no difficulty) to 3 (unable to do).
Correlation of SF36 and HAQ-DI results | through study completion, an average of 24 weeks
  Correlation of SF36 and HAQ-DI results. The HAQ-DI is a health assessment questionnaire - disability index that consists of 8 subcategories. For each the single scales range from 0 (no difficulty) to 3 (unable to do). SF36 is a 36 items short form health survey and consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Treatment satisfaction: TSQM-14 scores | at week 4
  Treatment Satisfaction Questionnaire for Medication (TSQM-14) scores. The TSQM items are answered on 5- or 7-point Likert type scale and cover four domains: effectiveness; side effects; convenience and global satisfaction. A score can be obtained for each domain by summing of the corresponding items transformed on a 0-100 scale; higher values indicate higher satisfaction, better perceived effectiveness, lower burden associated to side-effects, better convenience.
Treatment satisfaction: TSQM-14 scores | at week 12
  Treatment Satisfaction Questionnaire for Medication (TSQM-14) scores. The TSQM items are answered on 5- or 7-point Likert type scale and cover four domains: effectiveness; side effects; convenience and global satisfaction. A score can be obtained for each domain by summing of the corresponding items transformed on a 0-100 scale; higher values indicate higher satisfaction, better perceived effectiveness, lower burden associated to side-effects, better convenience.
Treatment satisfaction: TSQM-14 scores | at week 16
  Treatment Satisfaction Questionnaire for Medication (TSQM-14) scores. The TSQM items are answered on 5- or 7-point Likert type scale and cover four domains: effectiveness; side effects; convenience and global satisfaction. A score can be obtained for each domain by summing of the corresponding items transformed on a 0-100 scale; higher values indicate higher satisfaction, better perceived effectiveness, lower burden associated to side-effects, better convenience.
Treatment satisfaction: TSQM-14 scores | at week 24
  Treatment Satisfaction Questionnaire for Medication (TSQM-14) scores. The TSQM items are answered on 5- or 7-point Likert type scale and cover four domains: effectiveness; side effects; convenience and global satisfaction. A score can be obtained for each domain by summing of the corresponding items transformed on a 0-100 scale; higher values indicate higher satisfaction, better perceived effectiveness, lower burden associated to side-effects, better convenience.
Patient's expectation on treatment | at baseline
  Patient's expectation on treatment asked and documented as free text
Patient's expectation on treatment | at week 12
  Patient's expectation on treatment asked and documented as free text
Patient's expectation on treatment | at week 24
  Patient's expectation on treatment asked and documented as free text
Correlation of TSQM-14 results and patient's expectation on treatment | through study completion, an average of 24 weeks
  Correlation of TSQM-14 results and patient's expectation on treatment
drug accountability | at week 4
  Evaluation of results of treatment adherence (drug accountability) using patient diary
drug accountability | at week 12
  Evaluation of results of treatment adherence (drug accountability) using patient diary
drug accountability | at week 16
  Evaluation of results of treatment adherence (drug accountability) using patient diary
drug accountability | at week 20
  Evaluation of results of treatment adherence (drug accountability) using patient diary
drug accountability | at week 24
  Evaluation of results of treatment adherence (drug accountability) using patient diary
eGFR (estimated glomerular filtration rate) | at baseline
  eGFR value
eGFR (estimated glomerular filtration rate) | at week 4
  eGFR value
change in eGFR (estimated glomerular filtration rate) | at week 4
  eGFR change to BL
eGFR (estimated glomerular filtration rate) | at week 12
  eGFR value
change in eGFR (estimated glomerular filtration rate) | at week 12
  eGFR change to BL
change in eGFR (estimated glomerular filtration rate) | at week 16
  eGFR change to BL
eGFR (estimated glomerular filtration rate) | at week 16
  eGFR value
change in eGFR (estimated glomerular filtration rate) | at week 20
  eGFR change to BL
eGFR (estimated glomerular filtration rate) | at week 24
  eGFR value
change in eGFR (estimated glomerular filtration rate) | at week 24
  eGFR change to BL
blood pressure (mmHg) | at baseline
  blood pressure (mmHg) Systolic or Diastolic Blood Pressure
blood pressure (mmHg) | at week 4
  blood pressure (mmHg) Systolic or Diastolic Blood Pressure
change in blood pressure (mmHg) | at week 4
  blood pressure (mmHg) Systolic or Diastolic Blood Pressure change to BL
blood pressure (mmHg) | at week 12
  blood pressure (mmHg) Systolic or Diastolic Blood Pressure
change in blood pressure (mmHg) | at week 12
  blood pressure (mmHg) Systolic or Diastolic Blood Pressure change to BL
blood pressure (mmHg) | at week 16
  blood pressure (mmHg) Systolic or Diastolic Blood Pressure
change in blood pressure (mmHg) | at week 16
  blood pressure (mmHg) Systolic or Diastolic Blood Pressure change to BL
blood pressure (mmHg) | at week 20
  blood pressure (mmHg) Systolic or Diastolic Blood Pressure
change in blood pressure (mmHg) | at week 20
  blood pressure (mmHg) Systolic or Diastolic Blood Pressure change to BL
blood pressure (mmHg) | at week 24
  blood pressure (mmHg) Systolic or Diastolic Blood Pressure
change in blood pressure (mmHg) | at week 24
  blood pressure (mmHg) Systolic or Diastolic Blood Pressure change to BL
pain characteristics measured by QST (quantitative sensory testing) | at Baseline
  Correlation of pain characteristics measured by QST, VAS pain and pain relief
pain characteristics measured by QST (quantitative sensory testing) | at week 4
  Correlation of pain characteristics measured by QST, VAS pain and pain relief
pain characteristics measured by QST (quantitative sensory testing) | at week 8
  Correlation of pain characteristics measured by QST, VAS pain and pain relief
pain characteristics measured by QST (quantitative sensory testing) | at week 12
  Correlation of pain characteristics measured by QST, VAS pain and pain relief
pain characteristics measured by QST (quantitative sensory testing) | at week 24
  Correlation of pain characteristics measured by QST, VAS pain and pain relief
adverse events (AEs) | through study completion, an average of 24 weeks
  Documentation of type, frequency and seriousness of adverse events (AEs)
Infections | through study completion, an average of 24 weeks
  Incidence rates of serious infection events (SIEs),
Documentation of all lab abnormalities | through study completion, an average of 24 weeks
  incidence rates of lab abnormalities
Cardiovascular events | through study completion, an average of 24 weeks
  incidence rates of cardio vascular events
Malignencies | through study completion, an average of 24 weeks
  incidence rates of malignancies

CONTACTS AND LOCATIONS:
Overall Officials: Harald Burkhardt, MD, Principal Investigator — Fraunhofer IME
Locations (6):
- Germany (6):
  - Charité Universitätsmedizin Berlin, Med. Klinik mit Schwerpunkt Rheumatologie und klinische Immunologie, Berlin
  - Rheumatologische Schwerpunktpraxis im Ärztehaus am Walter-Schreiber-Platz, Berlin
  - CIRI - Centrum für innovative Diagnostik & Therapie, Rheumatologie/ Immunologie GmbH, Frankfurt
  - Katholische Kliniken Rhein-Ruhr, St. Elisabeth Gruppe GmbH, Rheumazentrum Ruhrgebiet, Herne
  - Praxis Prof. Dr. Kellner, München
  - Rheumazentrum Ratingen, Ratingen